CLINICAL TRIAL: NCT02473328
Title: Non-comparative Phase II Open Study Evaluating the Efficacy of a Reduced Dose Atazanavir / Ritonavir 200/100 mg + 2 NRTI in HIV-1-infected Patients With Virological Success With Atazanavir / Ritonavir 300/100 mg + 2 NRTI
Brief Title: Study Evaluating the Efficacy of a Reduced Dose Atazanavir in HIV-1-infected Patients
Acronym: ATALOW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Collaborators: INSERM UMR S 1136 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREPATS 003
Record Dates: First submitted 2015-05-27; First posted 2015-06-16 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: HIV-1 Infection
Keywords: dose reduction study
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non comparative open study (Experimental): In patients signed an informed consent and meeting all the eligibility criteria at the time of the run-in (S-4), switch of antiretroviral therapy Atazanavir 300 mg/ritonavir 100 mg once a day to Atazanavir 200 mg/ritonavir 100 mg once a day without changing the combination of 2 NRTIs associated.
  The administration will be done once a day orally for 48 weeks.
  Interventions: Drug: Atazanavir 200 mg/r

INTERVENTIONS:
Drug: Atazanavir 200 mg/r — 1. In patients signed an informed consent and meeting all the eligibility criteria at the time of the run-in (S-4),
  2. switch of antiretroviral therapy Atazanavir 300 mg/ritonavir 100 mg once a day to Atazanavir 200 mg/ritonavir 100 mg once a day without changing the combination of 2 NRTIs associated.
  The administration will be done once a day orally for 48 weeks.
  The usual recommended dose of atazanavir is 300 mg once daily with 100 mg of ritonavir once daily with food. Ritonavir acts by potentiating the pharmacokinetics of atazanavir.
  Other Names: ritonavir 100mg

SUMMARY:
The goal of antiretroviral therapy should be maintaining undetectable plasma viral load, only present condition to prevent the progression of the disease, improve immune restoration and prevent the emergence of viral resistance mutations. In addition to the individual benefit, antiretroviral treatment reduces the transmission of HIV from an infected person to sexual partners. There is to date no alternative strategy to antiretroviral treatment and antiretroviral therapy, even extended, does not allow viral eradication.

The need to maintain antiretroviral therapy for life raises the long-term safety concerns of it, even with the latest molecules. Also, one of the key issues in clinical research is whether after reaching undetectable viral load, antiretroviral treatment can be reduced in order to reduce exposure to molecules. Indeed, this treatment of "maintenance" could potentially need a smaller antiviral potency. On the other hand, reduction of antiretroviral treatment reduces costs, an important consideration in light of new global recommendations of treatment for all patients with T-cells CD4 below 500 / mm3.

The alleviation of antiretroviral therapy is to either reduce the number of molecules by making monotherapies or dual therapy, or to realize or intermittent treatment is to reduce the doses of molecules such as randomized ENCORE -1 showing the equivalence of a dose of Efavirenz 400mg instead of 600mg in naive patients.

Atalow study has the sense to lower the dose of Atazanavir / Ritonavir in combination with two NRTI to reduce exposure to this molecule and its cost while maintaining an undetectable viral load.

DETAILED DESCRIPTION:
Protease inhibitors (PIs) are key treatments in the current therapeutic strategy. They have major qualities such as their antiviral potency and high genetic barrier.

However, their long-term use is associated with gastrointestinal side effects, metabolic disorders (lipid, carbohydrate, lipohypertrophy) and cardiovascular comorbidities, renal and bone. The decrease in IP doses would reduce this predominantly concentration-dependent toxicity.

Atazanavir (Reyataz) was the first protease inhibitor once daily approved in 2003 for the treatment of HIV patients. Its favorable safety profile, ease of making and effectiveness have made treatment widely used and recommended first line. Atazanavir is recommended in Europe in naïve patient at the 300 mg dose once daily boosted with ritonavir 100 mg and in the pretreated patient at the 300 mg boosted with 100mg ritonavir or a dose of 400 no boosted mg in combination with two other antiretroviral drugs.

After oral administration, atazanavir is rapidly absorbed with improved variable bioavailability with food intake (40% increase in Cmin) and dependent on the gastric potential hydrogen (pH). Atazanavir is highly bound to plasma proteins (86%) and is largely metabolised by the isoform 3A4 (CYP3A4) cytochrome P450. There is great variability in the pharmacokinetics of atazanavir between patients due to inter-individual variability in the expression and function of CYP3A4. Co-administration of ritonavir increased 11.9 times Cmin and decreases the interindividual variability. The major effect of ritonavir is to decrease hepatic clearance of atazanavir. Its half-life of elimination is 8.6 hours when administered at 300 mg with 100 mg of ritonavir. 90% inhibitory concentration of atazanavir adjusted to the plasma protein binding (PBA EC90) is 14ng / ml. At the standard dose of 300 mg taken with 100 mg ritonavir once daily, the mean trough concentration at steady state is according to research from 526 ng / ml and 862 ng / ml in HIV patients. Residual therapeutic levels (Cmin) must be greater than 150 ng / ml. The relationship between the residual plasma concentrations and virologic response was demonstrated in the naive patient pharmacokinetic substudy BMS 089.

If the inhibitor atazanavir is best tolerated on lipid map protease is responsible for specific side effects such as hyperbilirubinemia and nephrolithiasis, concentration-dependent side effects. Indeed, atazanavir is responsible for a reversible elevation of unconjugated bilirubin, inhibiting glucuronide conjugation bilirubin by UGT1A1. This effect, not easily concealed by the patient, is an important and annoying side effects that may interfere with treatment adherence. This hyperbilirubinemia is concentration-dependent, with elevated bilirubin most common grade 3-4, atazanavir C min is greater than 760 ng / ml (600 to 850 ng / ml according to studies).

No boosted atazanavir may be used but with caution. Indeed, its use should be avoided in patients with a history of failure or virological resistance mutations in a patient with poor adherence and in patients taking other drugs that could interfere with atazanavir. Pharmacokinetic studies at a dose of 400 mg without ritonavir showed a concentration below the expected minimum concentration of 150 mg / l in 60% of cases. In addition, the use of no boosted atazanavir with tenofovir has been little studied and requires close monitoring pharmacological given the interaction between these two molecules (decrease of approximately 25% of the concentration of atazanavir when without ritonavir in combination with tenofovir. Finally, in the INDUMA study, there was no virologic rebounds in this strategy.

Monotherapy atazanavir is not recommended in light of studies showing virological failures under this strategy.

The evaluation of atazanavir / r 200/100 in healthy patient presented at CROI meeting in 2001 in Phase II studies showed a mean Cmin 378 ng / ml (SD = 286 EC).

A retrospective cohort study in 14 Thai patients with virologic success in switched to atazanavir / r 200/100 showed maintenance of a CV less than 50 copies / ml over a median follow-up 68 weeks (range 12-165 weeks). Five of the patients had a dose of atazanavir Cmin had greater than 150 ng / ml (mean Cmin = 572 ng / ml). The lipid profile was improved but not significantly.

A pharmacokinetic study of 22 Thai patients on atazanavir / r 300/100 in switched to atazanavir / r 200/100 2 NRTIs showed minimum concentrations reduced by 48.6% remaining above the minimum therapeutic concentration of 150 ng / ml (mean Cmin = 700 ng / ml EC = 470).

A case study conducted in 14 Italian patients (10 Caucasian and 4 of African origin) with virologic suppression (CV below 50 copies / ml) with atazanavir / r 300/100 mg + 2 NRTI showed a maintenance of viral efficacy after the switch to atazanavir / r 200/100 on a 1 year average follow-up. Atazanavir C min was above Cmin for all except 2 patients (whose viral load remained below 50 copies / ml), with a mean Cmin 713ng / ml. Bilirubin decreased after the switch.

Recently, a pharmacokinetic simulation study was performed in a majority of Caucasian patients for atazanavir / r doses at 300/50 mg, 200/50 mg and 200/100 mg. The lowest concentrations of atazanavir after dose reduction 200/100 averaged 520 ng / ml (EC = 448) and all remained above the recommended Cmin.

In total, these four dose reduction studies of atazanavir / r 200/100 in treatment-experienced patients with virologic average Cmin were between 520 and 713ng / ml, well above the therapeutic Cmin.

The decrease in atazanavir dose showed a significant decrease of serum bilirubin 14.88μmol / l after 2 weeks.

This test is within the overall reflection optimization of antiretroviral therapy.

In view of the existing data of Pharmacology and few data Italian and Thai in switched patients to atazanavir / r 200/100 mg, the ATALOW study hypothesizes that a lower dose of atazanavir / r 200 / 100 mg is able to maintain an undetectable viral load in treatment-experienced patients with virologic success.

The expected benefits of the reduction in the dose of atazanavir / r 200/100 mg + would be:

* A better tolerance especially in terms of bilirubin
* A more robust strategy that using no boosted atazanavir with the possibility of using tenofovir in combination NRTI.
* The same simplicity taking once a day
* Reduced costs (2,730 euros less per patient per year).

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection.
* Age ≥ 18 years
* Plasma HIV-RNA level ≤ 50 copies/mL during the last 24 months prior to screening visit (W-4), documented by at least 4 time-points
* Stable antiretroviral treatment with 2 NRTI + ATV/r 300/100 for at least 6 month
* CD4+ lymphocytes > 300 cells/mm3
* Negative urinary pregnancy test and use of efficient contraception for women of childbearing potential
* Signed informed consent
* Patient affiliated or beneficiary of a national insurance scheme (article L1121-11 of the Public health code) (the Medical aid of State or SOUL is not a national insurance scheme)

Exclusion Criteria:

* HIV-2 infection.
* Patient with resistant mutation for ATV and/or NRTI used on the available genotypic test
* Concomitant treatment using one or more molecules interacting with hepatic cytochromes
* Ongoing cancer. Patients with cancer considered cured for at least six months may be included.
* Active viral hepatitis C requiring a specific treatment during the 48 weeks of the trial
* hemodialysis patients
* Pregnant women, breastfeeding women or women wishing to be pregnant during the study period
* Patient with a history of non-compliance or irregular follow-up
* Subjects under "Backup justice" (judicial protection due to temporarily and slightly diminished mental or physical faculties), or under legal guardianship
* Subjects participating in another clinical trial evaluating different therapies and including an exclusion period that is still in force during the screening phase
* All conditions (use of alcohol, drugs, etc.) judged by the investigator to possibly interfere with trial protocol compliance, adherence and/or trial treatment tolerance
* Non-attendance which could impede the trial participation (travel abroad, moving, impending transfer...)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Measure of effectiveness assessed by maintaining undetectable plasma HIV viral load (viral load ≤ 50 copies / ml) during the all period of this study of treatment with ATV / r 200/100 mg + 2 NRTIs, for all patients. | one year
Measure of safety (adverse events) | one year
  Number of participant with adverse events
Measure of tolerability assessed by number of patient interrupting the study treatment for virological failure | one year
Measure of effectiveness assessed by number of patient maintaining a target trough plasma concentration of atazanavir associated to efficacy: | one year
  Residual plasma concentrations of ATV / r (Dates and last dose of antiretroviral schedules and the association or not with food ) will be performed at day 0 before changing dose reduction of atazanavir, week 12 and week 24 for all patients.
Measure of effectiveness assessed in patient with virological failure number of patient dysplaing HIV strains with mutations associated to treatment resistance | one year
Measure of tolerability assessed by number of patient interrupting the study treatment for in tolerance | one year
Measure of tolerability assessed by quantification of bilirubinemia | one year
Measure of tolerability assessed by quantification of creatininemia | one year

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière; Claudine Duvivier, MD, Principal Investigator — Hôpital Necker-Enfants Malades; Yazdan Yazdanpanah, MD, Principal Investigator — Groupe hospitalier Bichat-Claude Bernard
Locations (1):
- DUDOIT Yasmine, Paris, France